CLINICAL TRIAL: NCT03423030
Title: Safety, Tolerability, Pharmacokinetic Profile and Ex-vivo Antitubercular Activity of PBTZ169 Formulated as Spray- Dried Dispersion Versus Native Crystal Powder: Single Ascending Doses, Randomized, Placebo- Controlled, Cross-over Phase Ia Trial in Healthy Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Ex-vivo Antitubercular Activity of PBTZ169 Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovative Medicines for Tuberculosis (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IM-006-11
Record Dates: First submitted 2018-01-24; First posted 2018-02-06 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Panel A - Active (Experimental): N = 6, 10 mg then 40 mg of PBTZ169 Formulation
  Interventions: Drug: PBTZ169 Formulation
- Panel A - Placebo (Placebo Comparator): N = 2, 10 mg then 40 mg of matching placebo
  Interventions: Drug: Placebo
- Panel B - Active (Experimental): N = 6, 20 mg then 80 mg of PBTZ169 Formulation
  Interventions: Drug: PBTZ169 Formulation
- Panel B - Placebo (Placebo Comparator): N = 2, 20 mg then 80 mg of matching placebo
  Interventions: Drug: Placebo
- Panel C - Active (Experimental): N = 6, First dosing of Panel C with 160 mg PBTZ169 Formulation then Second dosing of Panel C with 160 mg PBTZ169 Native Crystalline Powder (NCP)
  Interventions: Drug: PBTZ169 Formulation; Drug: PBTZ169 NCP
- Panel C - Placebo (Active Comparator): N = 2, 160 mg of matching placebo for the two interventions
  Interventions: Drug: Placebo
- Panel D - Active (Experimental): N = 6, First dosing of Panel D with 320 mg PBTZ169 Formulation then Second dosing of Panel D with 320 mg PBTZ169 Native Crystalline Powder (NCP)
  Interventions: Drug: PBTZ169 Formulation; Drug: PBTZ169 NCP
- Panel D - Placebo (Active Comparator): N = 2, 320 mg of matching placebo for the two interventions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBTZ169 Formulation — PBTZ169 Formulation supplied as powder for oral solution
  Arms: Panel A - Active; Panel B - Active; Panel C - Active; Panel D - Active
Drug: Placebo — matching placebo supplied as powder for oral solution
  Arms: Panel A - Placebo; Panel B - Placebo; Panel C - Placebo; Panel D - Placebo
Drug: PBTZ169 NCP — PBTZ169 NCP supplied as powder for oral solution
  Arms: Panel C - Active; Panel D - Active

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose study conducted at one study center in Switzerland.

Four (4) panels (A, B, C and D) of 8 male subjects (6 active and 2 placebo) each undergoing 2 investigation periods and receiving either single doses of PBTZ169 at increasing dose levels or a matching placebo.

Subjects will participate in only one panel. Blocks of 4 subjects (3 under active treatment, 1 under placebo) will be investigated in parallel. Panels A and B are interleaved.

Safety will be assessed throughout the study; serial ECGs and serial blood samples will be collected for the safety and PK assessment of PBTZ169.

Dose escalation will be allowed once the Trial Safety Board has determined that adequate safety and tolerability after panel B and panel C completion has been demonstrated to permit proceeding to the next panel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged between 18 and 48 years
* Body weight (BW) ranging between 55 and 95 kg, providing body mass index (BMI) is between 18 and 28 kg/m2
* Absence of significant findings in the medical history and physical examination as judged by the Investigator, especially for cardiovascular, pulmonary, haematological and nervous systems
* Absence of significant laboratory abnormalities as judged by the Investigator. Gilbert's syndrome (increased total and unconjugated bilirubin when fasting) will be accepted if mild
* Absence of clinically significant abnormalities on 12-lead ECG
* Negative urine drug screen (amphetamines, benzodiazepines, cannabis, cocaine, opiates)
* Commitment to refrain from travel outside Europe over the whole study duration
* Ability to understand the procedures, agreement to participate and willingness to give written informed consent
* Co-operative attitude and availability for scheduled visits over the entire study period

Exclusion Criteria:

* History of major cardiovascular, pulmonary, hepatic, immunological, renal, haematological, gastrointestinal, genitourinary, neurological, or rheumatologic disorders
* Active diseases of any type, including inflammatory disorders and infections. Mild acne is permissible providing no systemic or local treatment is provided or planned (except for cleaning lotions)
* History of significant allergy or asthma. Allergic rhinitis or conjunctivitis is acceptable if non-symptomatic when starting the study and if symptoms are not anticipated to occur during the study to a point that would require corticosteroid therapy (e.g. in case of annual use)
* History of cardiovascular dysfunction if considered as clinically relevant (conduction abnormality, arrhythmia, bradycardia, angina pectoris, cardiac hypertrophy unless elicited by training, pulmonary embolism)
* Hypertension defined as supine blood pressure >150/90 mmHg or recurrent hypotensive events considered as clinically relevant or documented orthostatic hypotension
* Sick sinus syndrome, known long QT syndrome, reproducible observation of QTc ≥ 440 msec or of pronounced sinus bradycardia (<40 bpm/min)
* Intense sport activities. Moderate sport is acceptable and activities should remain fairly constant throughout the study
* Any clinically significant laboratory values on screening that are not within normal range on single repeat (Gilbert's syndrome acceptable if mild)
* Positive hepatitis B and C antigen screen
* Positive HIV antibody screen or screen not performed
* Any recent acute illness or sequelae thereof which could expose the subject to a higher risk or might confound the results of the study
* Treatment in the previous three months with any drug known to have well-defined potential for toxicity to a major organ
* History of hypersensitivity to any drug if considered as serious
* Use of any medication the week prior to study or as based on the 5 plasma half-life rule and throughout study, including aspirin or other over-the-counter (OTC) preparations. Paracetamol is permissible before and during the study as a rescue medication but only with Investigator's permission
* Participation in a clinical investigation or blood donation of 500 ml within the past 3 months
* History of relevant alcohol or drug abuse
* Usual smoking during the last month before participation in the study. Consumption of ≤ 5 cigarettes/day or equivalent is acceptable providing the subject can totally refrain from smoking from one week before and during the whole study duration
* Usual consumption of a large quantity of coffee, tea, chocolate (more than 4 cups/day) or equivalent (Cola drinks), during the last month before participation in the study
* Current regular (i.e. 3 times per week or more) consumption of large quantities of alcohol or wine (>0.5 L wine/day) or equivalent (i.e. more than 35 g ethanol per day), during the last month before participation in the study
* Project to conceive a child during the study period (by principle of precaution, while no indication exists for a definite reproductive risk following paternal exposure)
* Psychological status which could impact on the subject's ability to give informed consent
* Any feature of the subject's medical history or present condition which, in the Investigator's opinion, could confound the results of the study, complicate its interpretation, or represent a potential risk for the subject

Ages: 18 Years to 48 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of increasing single oral doses of PBTZ169 Formulation in healthy male adult subjects evaluated by Treatment Emergent Adverse Events (TEAEs). | Days 0-17
  Evaluation by thorough monitoring of Treatment Emergent Adverse Events (TEAEs) following doses of PBTZ169 Formulation, PBTZ169 NCP or placebo

SECONDARY OUTCOMES:
Relative oral bioavailability assessment of the PBTZ169 Formulation in comparison to NCP in healthy male subjects | Days 0-2
  Estimation from the ratio of area under plasma concentration curves (AUCs) determined after the administration of each formulation
Pharmacokinetics (PK) of single oral doses of PBTZ169 using Cmax | Days 0-2
  Determination of non-compartmental PK parameter Maximum Plasma Concentration [Cmax] after determination of the amount of the parent compound and its known metabolites in plasma samples
Pharmacokinetics (PK) of single oral doses of PBTZ169 using Tmax | Days 0-2
  Determination of non-compartmental PK parameter Time of maximum observed Plasma Concentration [Tmax] after determination of the amount of the parent compound and its known metabolites in plasma samples
Pharmacodynamics (PD) exploration after single oral doses of PBTZ169 Formulation and NCP | Days 0-1
  Determination of ex-vivo antitubercular activity of serum samples obtained from subjects
Broncho-alveolar passage exploration after single oral doses of PBTZ169 Formulation and NCP (tentative) | Days 0-1
  PBTZ169 concentrations in sputum samples collected by hypertonic NaCl-induction

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland